CLINICAL TRIAL: NCT04548960
Title: Molecular Profiles Associated With Resistance Development in Cancer Patients. Prospective Exploratory Study From 3 Cancer Locations: TNBC or Locally Advanced or Metastatic, Non-small Cell or Pancreatic or Bronchial Cancers
Brief Title: OncoSNIPE - Study of Molecular Profiles Associated With the Development of Resistance in Solid Cancer Patients
Acronym: OncoSNIPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oncodesign SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A02018-45
Record Dates: First submitted 2020-07-06; First posted 2020-09-16 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2020-09

CONDITIONS: CANCER
Keywords: Resistance; Markers; Exome; Transriptome; Immunological Profil
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study a part of samples (blood and biopsies) will be collected specifically for this study. This is why the study is therefore interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cancer patients (Other): cancer patients To explore the phenomena of resistance during the therapeutic response and/or the progression of the pathology, the investigatorswill used a multidisciplinary approach including high-throughput sequencing (Exome-seq and RNAseq) from blood and tumor samples and immunological profil by ELISA
  Interventions: Other: cancer patients

INTERVENTIONS:
Other: cancer patients — Blood sample RNA_seq at time of diagnostic, best response and relapse ; Biopsy Exom_seq and RNA_seq at time of diagnostic and relapse Immulogical Profiling at time of diagnostic, best response and relapse

SUMMARY:
Precision medicine is considered to be one of the major issues in patient care. A lot of research has already proven itself with the implementation of targeted therapies including immunotherapies offering patients improved response and survival rates. But despite these major therapeutic advances, resistance to anti-cancer treatment is a major obstacle in the care of patients. Indeed, to date, many patients die of cancer, 9.6 million deaths worldwide in 2018. Nowadays, improving understanding of the mechanisms of resistance of cancer cells to anti-tumor treatments is therefore a major issue. The great diversity of molecular mechanisms involved in the phenomena of resistance to treatment, whether intrinsic (de novo, or primary) or acquired (secondary), constitutes a real therapeutic challenge. Indeed, a better understanding of the mechanisms of resistance would make it possible to explore new therapeutic strategies making it possible to circumvent these phenomena of escape in different types of cancer. It is in this context that the OncoSNIPE project was developed. The objective of this project is to identify early and / or late markers of resistance to treatment in 3 different pathologies concerned with resistance issues: triple negative breast cancer or Lum B or locally advanced or metastatic non -small-cell lung cancer or pancreatic cancer. In this project, in order to best cover the diversity of mechanisms involved in these resistances, the investigators propose a multidisciplinary approach with clinical, genomic, transcriptomic and immunological dimensions of the pathology through the data collected from 600 patients (200 for each pathology) for 4 years

DETAILED DESCRIPTION:
Precision medicine is considered to be one of the major issues in patient care. A lot of research has already proven itself with the implementation of targeted therapies including immunotherapies offering patients improved response and survival rates. But despite these major therapeutic advances, resistance to anti-cancer treatment is a major obstacle in the care of patients. Indeed, to date, many patients die of cancer, 9.6 million deaths worldwide in 2018. Nowadays, improving understanding of the mechanisms of resistance of cancer cells to anti-tumor treatments is therefore a major issue. The great diversity of molecular mechanisms involved in the phenomena of resistance to treatment, whether intrinsic (de novo, or primary) or acquired (secondary), constitutes a real therapeutic challenge. Indeed, a better understanding of the mechanisms of resistance would make it possible to explore new therapeutic strategies making it possible to circumvent these phenomena of escape in different types of cancer. It is in this context that the OncoSNIPE project was developed. The objective of this project is to identify early and / or late markers of resistance to treatment in 3 different pathologies concerned with resistance issues : triple negative breast cancer or lum B or locally advanced or metastatic non- small-cell lung cancer or pancreatic cancer. In this project, in order to best cover the diversity of mechanisms involved in these resistances, the investigators propose a multidisciplinary approach with clinical, genomic, transcriptomic and immunological dimensions of the pathology through the data collected from 600 patients (200 for each pathology) for 4 years.

The patient populations targeted in this study have one common thing: rapid progression of their pathology, making it possible to obtain models for evaluating markers of early and / or late responses over the period of follow-up of 2-year post-inclusion patients, and thus provide the information necessary to understand the resistance mechanisms.

To explore the phenomena of resistance, during the therapeutic response and / or the progression of the pathology, the investigators will used a multidisciplinary approach including high-throughput sequencing (Exome-seq and RNAseq) and immunological profil by ELISA . Patients will have long-term follow-up with different biological samples, at baseline (blood and biopsy) and at each tumoral evaluation or tumoral progression evaluated by medical imaging.

ELIGIBILITY:
Inclusion Criteria:

1. General

   * Adult patient, 18 years of age or older
   * Naive chemo patient
   * Performant status: 0,1 or 2.
   * Life expectancy> 3 months
   * Subject affiliated to a social security and health insurance scheme
   * Subject having dated and signed informed consent
   * For women of childbearing age (negative pregnancy test): effective contraception
2. Pancreatic cancer:

   * Patient receiving a biopsy, as part of the usual care of the patient:

     * Either from the primary tumor
     * Either a metastasis for a strong suspicion of locally advanced or metastatic pancreatic ductal adenocarcinoma;
   * With advanced or metastatic tumors (liver, lungs, peritoneum, others) that cannot benefit from local or locoregional treatment;
   * Presence of target lesion (s) measurable according to RECIST criteria
   * Patient who cannot be treated by surgery or radiotherapy
3. Lung cancer:

   * Patient with histologically proven non-small cell lung cancer
   * Locally advanced stage IIIB or IV
   * Treatment with chemotherapy, targeted therapy, immunotherapy
   * Tissue available after analysis of the usual biomarkers in the event of a non-epidermoid tumor
   * Rate of tumor cells observed on biopsies must be ≥ 30%.
   * Presence of measurable target lesion or disease assessable according to RECIST criteria
4. Breast cancer:

   * Breast cancer of recent diagnosis, histologically proven.
   * Triple negative breast cancer: negativity of estrogen and progesterone receptors in the tumor (<10%), absence of HER2 overexpression according to the IHC classification (score 0 or 1+) and / or FISH negative
   * or
   * LumB: RO positive, RP positive or negative, HER2 negative, high proliferation;
   * Stage I to III for triple negative breast cancer (including stage T4d = inflammatory cancer), Stage II or III of the UICC classification for LumB
   * Non-metastatic patient (M0 according to TNM classification)
   * Rate of tumor cells observed on biopsies must be ≥ 30%
   * Patient who cannot be treated exclusively by surgery or radiotherapy

Exclusion Criteria:

General

* History of chemotherapy (except adjuvant completed for more than at least 6 months) or radiotherapy
* Patient whose monitoring and treatment will not be carried out in the study health establishments;
* Tumor not histologically proven;
* Life expectancy of less than 3 months
* Pregnancy or breastfeeding
* Refusal to participate in the trial
* Persons deprived of their liberty, persons under guardianship or curatorship
* Inability to submit to the medical follow-up of the test for social or psychological reasons
* No affiliation to a social security scheme or state medical aid (AME) or universal medical coverage (CMU)
* Any condition for which participation in the protocol would present a risk or which would not make it possible to comply with the requirements of the protocol according to the investigator
* History of other cancers in the last 5 years except cervical cancer and skin cancer of the basal or epidermoid cells treated
* Known HIV seropositivity Specific

Pancreatic cancer:

* Other histologies: neuroendocrine cancer, acinar cancer, pancreatic metastasis of another cancer
* Patient who cannot benefit from chemotherapy (Performans status (PS) 3 - 4);
* Other progressive cancer during the management of pancreatic cancer;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-01-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Combinatory analysis of genomic, transcriptomic and immunological profile | up to 24 months
  1. Genomic changes associated with early and/or late resistance to treatment given alone or in combination in patients [ Time Frame: Through study completion, up to 2 years ]
  2. Transcriptomic changes associated with early and/or late resistance to treatment given alone or in combination in patients [ Time Frame: Through study completion, up to 2 years ]
  3. Immunophenotypic changes associated with early and/or late resistance to treatment given alone or in combination in patients [ Time Frame: Through study completion, up to 2 years ]

SECONDARY OUTCOMES:
Progression-free survival | up to 24 months
  Clinical data from Baseline until 24 months
Over Survival | up to 24 months
  Clinical data from Baseline until 24 months

CONTACTS AND LOCATIONS:
Overall Officials: FRANCOIS GHIRINGHELLI, MD, Principal Investigator — Centre Georges François Leclerc
Locations (11):
- France (11):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Chu de Besancon, Besançon, Bourgogne-Franche-Comté
  - CGFL, Dijon, Bourgogne-Franche-Comté
  - Chu Dijon Bourgogne, Dijon, Bourgogne-Franche-Comté
  - Institut de Cancerologie de Lorraine, Nancy, Grand Est
  - Institut Godinot, Reims, Grand Est
  - Hopitaux Universitaires de Strasbourg, Strasbourg, Grand Est
  - Chu de Poitiers, Poitiers, Nouvelle-Aquitaine
  - Institut Paoli Calmettes, Marseille, PACA
  - APHP - Hôpital Beaujon, Clichy, Paris
  - Institut Curie, Paris

REFERENCES:
- [Derived] Vachenc S, Gobbo J, Moujarrebe SE, Desmoulins I, Gilabert M, Beau-Faller M, Mitry E, Girard N, Bertaut A, Dusetti N, Iovanna JL, Yousfi R, Pierrat F, Bruno R, Cueff A, Boidot R, Genne P. OncoSNIPE(R) Study Protocol, a study of molecular profiles associated with development of resistance in solid cancer patients. BMC Cancer. 2022 Jan 6;22(1):41. doi: 10.1186/s12885-021-09134-3. PMID 34991520
- See also: OncoSNIPE Program description — https://www.oncodesign.com/en/our-technologies/oncosnipe-technology